CLINICAL TRIAL: NCT06585241
Title: A Phase 3b/4, Open-label Study to Assess the Immunogenicity and Safety of mRNA COVID-19 Variant-containing Vaccine Formulations
Brief Title: A Study to Investigate the Immunogenicity and Safety of mRNA COVID-19 Variant-containing Vaccine Formulations
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-1273-P403
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Variant; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a Phase 3b/4 open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA-1273 Variant-containing Formulation (Experimental): Participants will receive an intramuscular (IM) injection of a mRNA-1273 variant-containing formulation (mRNA-1273.167, mRNA-1273.712, or mRNA-1273.251).
  Interventions: Biological: mRNA-1273 Variant-containing Formulation

INTERVENTIONS:
Biological: mRNA-1273 Variant-containing Formulation — Sterile liquid for injection

SUMMARY:
The purpose of this study is to investigate the immunogenicity of mRNA COVID-19 variant-containing vaccine formulations against the vaccine matched variants and newly emerged variants of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

DETAILED DESCRIPTION:
This study uses a master protocol with a generic study design to allow flexibility in evaluating immunogenicity of variant-containing formulations of the mRNA-1273 COVID-19 vaccine. As different variant-containing vaccine formulations will be evaluated, each study intervention will be described in the subprotocol. For each evaluation of an updated variant vaccine, a new subprotocol will be generated.

ELIGIBILITY:
Key Inclusion Criteria:

* mRNA-1273.167 and mRNA-1273.712: Previously vaccinated adults aged ≥18 years
* mRNA-1273.251: Participants ≥65 years or ≥12 to <65 years of age with at least 1 risk factor for severe outcomes from COVID-19.
* Able to comply with study procedures based on the assessment of the Investigator.
* Female participants of childbearing potential may be enrolled in the study if the participant fulfills all the following criteria:

  * Has a negative pregnancy test at the Screening Visit and on the day of vaccination prior to vaccine dose being administered on Day 1.
  * Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose.
  * Has agreed to continue adequate contraception through 28 days following vaccine administration.

Key Exclusion Criteria:

* History of SARS-CoV-2 infection within 3 months prior to enrollment for mRNA-1273.167 and mRNA-1273.712 or within 6 months prior to enrollment for mRNA-1273.251.
* Is acutely ill or febrile (temperature 38.0°Celsius/100.4°Fahrenheit) less than 72 hours prior to or at the Screening Visit or Day 1. Participants meeting this criterion may be rescheduled within the Screening window.
* History of a diagnosis or condition that, in the judgment of the Investigator, is clinically unstable, or may affect participant safety, assessment of study endpoints, assessment of immune response, or adherence to study procedures.
* History of anaphylaxis or severe hypersensitivity reaction requiring medical intervention after receipt of any mRNA vaccine or therapeutic or any components of an mRNA vaccine or therapeutic.
* Receipt of COVID-19 vaccine within 3 months prior to enrollment for mRNA-1273.167 and mRNA-1273.712 or within 6 months prior to enrollment for mRNA-1273.251.
* Receipt of any licensed non-COVID-19 vaccine within 28 days before or planned receipt within 28 days after the study intervention, except an influenza vaccine, which may be given 14 days before or after receipt of the study intervention.
* Receipt of systemic immunosuppressants or immune-modifying drugs for >14 days total (within 6 months prior to Screening for mRNA-1273.167 and mRNA-1273.712 or within 180 days prior to Screening for mRNA-1273.251) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Receipt of systemic immunoglobulins or blood products (within 3 months prior to Screening for mRNA-1273.167 and mRNA-1273.712 or within 90 days prior to the Screening for mRNA-1273.251) or plans for receipt during the study.
* Has donated ≥450 milliliters of blood products within 28 days prior to the Screening Visit or plans to donate blood products during the study.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 764 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
mRNA-1273.167, mRNA-1273.712, and mRNA-1273.251 (Part A): Geometric Mean Value of Neutralizing Antibody Against COVID-19 Variants | Day 29
mRNA-1273.167, mRNA-1273.712, and mRNA-1273.251 (Parts A and B): Geometric Mean Fold Rise of Neutralizing Antibody Against COVID-19 Variants | Day 29
mRNA-1273.251 (Part A): Seroresponse Rate | Day 29

SECONDARY OUTCOMES:
mRNA-1273.251 (Part B): Geometric Mean Titer of Neutralizing Antibody Against COVID-19 Variants of Participants ≥12 to <65 Years Old and ≥65 Years Old | Day 29
mRNA-1273.167, mRNA-1273.712, and mRNA-1273.251 (Part A): Number of Participants with Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Study Withdrawal, and AEs of Special Interest | Day 1 through Day 29
mRNA-1273.251 (Part B): Number of Participants with Solicited Local and Systemic Adverse Reactions | Day 1 through Day 7
mRNA-1273.251 (Part B): Number of Participants with Unsolicited AEs | Day 1 through 28 days
mRNA-1273.251 (Part B): Number of Participants with SAEs, AEs of Special Interest, and AEs Leading to Study Withdrawal | Day 1 through Day 181

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - CenExel, Atlanta, Georgia
  - CenExel, Decatur, Georgia
  - Velocity Clinical Research, Baton Rouge, Louisiana
  - Velocity Clinical Research, Gulfport, Mississippi
  - Velocity Clinical Research, Omaha, Nebraska